CLINICAL TRIAL: NCT03219216
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Glecaprevir (GLE)/Pibrentasvir (PIB) in Treatment-Naïve Adults in Brazil With Chronic Hepatitis C Virus (HCV) Genotype 1 - 6 Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of Glecaprevir (GLE)/Pibrentasvir (PIB) in Treatment-Naive Adults in Brazil With Chronic Hepatitis C Virus (HCV) Genotype 1 - 6 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-156
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Virus (HCV); Genotype 1 - 6; Metavir System Fibrosis Score; Glecaprevir; Pibrentasvir; Treatment naïve; Cirrhosis; Compensated cirrhosis
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Fibrosis | interventions — glecaprevir and pibrentasvir; glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 weeks (Experimental): Arm A: Hepatitis C virus (HCV) genotype (GT) 1 to GT6 participants without cirrhosis (fibrosis stage F2 to F3) received glecaprevir (GLE)/pibrentasvir (PIB) 300 mg/120 mg once daily (QD) for 8 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir
- Arm B: GLE/PIB for 12 Weeks (Experimental): Arm B: HCV GT1 to GT6 participants with compensated cirrhosis (F4) received GLE/PIB 300 mg/120 mg QD for 12 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Film-coated tablet
  Other Names: ABT-493; ABT-530; MAVYRET

SUMMARY:
This was a Phase 3, open-label, multicenter study to evaluate the efficacy and safety of glecaprevir (GLE)/pibrentasvir (PIB) for an 8 or 12-week treatment duration in adults in Brazil with chronic hepatitis C virus (HCV) genotype (GT) 1 to GT6 infection, without cirrhosis or with compensated cirrhosis, who were HCV treatment-naïve.

DETAILED DESCRIPTION:
This was a Phase 3, open-label, multicenter study to evaluate the efficacy and safety of GLE/PIB for an 8- or 12-week treatment duration in adults in Brazil with chronic HCV GT1 to GT6 infection, without cirrhosis or with compensated cirrhosis with a METAVIR System Fibrosis Score of F2 to F3 (without cirrhosis) or F4 (with compensated cirrhosis) or equivalent, who were HCV treatment-naïve.

ELIGIBILITY:
Inclusion Criteria:

* Participant had positive plasma hepatitis C virus (HCV) antibody and HCV ribonucleic acid (RNA) viral load greater than or equal to 1000 IU/mL at Screening Visit.
* Participant must have been documented as without cirrhosis with METAVIR equivalent fibrosis stage of F2 to F3 or with compensated cirrhosis (F4) based on results of a liver biopsy, or FibroScan, or FibroTest score.
* Participants who were known to be HCV/Human Immunodeficiency Virus (HIV) co-infected may have been enrolled if they had a positive test result for anti-HIV antibody at Screening and were: naïve to treatment with any antiretroviral therapy (ART), or on a stable, qualifying HIV ART regimen for at least 8 weeks prior to Baseline.
* Participants with compensated cirrhosis only: Absence of hepatocellular carcinoma (HCC) within 3 months prior to Screening or a negative ultrasound at Screening.

Exclusion Criteria:

* Current hepatitis B virus (HBV) infection on screening tests.
* Any current or past clinical evidence of Child-Pugh B or C classification (score of > 6) or clinical history of liver decompensation including ascites on physical exam, including hepatic encephalopathy or variceal bleeding.
* Receipt of any investigational or commercially available anti-HCV agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (14):
- Brazil (14):
  - Hospital Universitário Cassiano Antônio Moraes - HCUFES /ID# 163512, Vitória, Espírito Santo
  - Hospital Universitario da Universidade Federal do Maranhao - CEPEC /ID# 163169, São Luís, Maranhão
  - Universidade Estadual de Maringá /ID# 166436, Maringá, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 163166, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre /ID# 163167, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles /ID# 163171, Porto Alegre, Rio Grande do Sul
  - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu /ID# 163066, Botucatu, São Paulo
  - Instituto de Infectologia Campinas /ID# 163175, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP /ID# 163054, Ribeirão Preto, São Paulo
  - Instituto de Infectologia Emilio Ribas /ID# 163170, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HC /ID# 163168, São Paulo, São Paulo
  - UNIFESP/Unidade de Atendimento Pesquisa Clínica 1 /ID# 164188, São Paulo
  - Centro de Referência e Treinamento DST/AIDS /ID# 163174, São Paulo
  - Hospital Heliopolis /ID# 163063, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Brown RS Jr, Collins MA, Strasser SI, Emmett A, Topp AS, Burroughs M, Ferreira R, Feld JJ. Efficacy and Safety of 8- or 12 Weeks of Glecaprevir/Pibrentasvir in Patients with Evidence of Portal Hypertension. Infect Dis Ther. 2022 Apr;11(2):913-924. doi: 10.1007/s40121-022-00599-8. Epub 2022 Feb 17. PMID 35174470
- [Derived] Peribanez-Gonzalez M, Cheinquer H, Rodrigues L, Lima MP, Alvares-da-Silva MR, Madruga J, Parise ER, Pessoa MG, Furtado J, Villanova M, Ferreira A, Mazzoleni F, Nascimento E, Silva GF, Fredrick L, Krishnan P, Burroughs M, Reuter T. Efficacy and safety of glecaprevir/pibrentasvir in treatment-naive adults with chronic hepatitis C virus genotypes 1-6 in Brazil. Ann Hepatol. 2021 Jan-Feb;20:100257. doi: 10.1016/j.aohep.2020.09.002. Epub 2020 Sep 17. PMID 32949786

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants were enrolled and received ≥ 1 dose of study drug.
Period: Overall Study
Arm/Group | Arm A: Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks | Arm B: GLE/PIB for 12 Weeks
Started | 75 | 25
Completed | 75 | 24
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Arm B: GLE/PIB for 12 Weeks: Arm B: HCV GT1 to GT6 participants with compensated cirrhosis (F4) received GLE/PIB 300 mg/120 mg once daily (QD) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm A: Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 Weeks | Arm B: GLE/PIB for 12 Weeks | Total
Number analyzed (Participants) | 75 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.87 (11.28) | 56.44 (9.62) | 54.51 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 5 | 36
  Male | 44 | 20 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White | 46 | 17 | 63
  Black or African American | 22 | 4 | 26
  Asian | 1 | 1 | 2
  Multi-race | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; less than 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last dose of study drug (week 20 or 24 depending on treatment regimen)
Population: All enrolled participants who received at least one dose of study drug. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders. Data are reported for the overall study population according to the prespecified analysis plan for this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: Glecaprevir (GLE)/Pibrentasvir (PIB) for 8 or 12 weeks
Arm/Group | All Participants
Number analyzed (Participants) | 100
percentage of participants | 98.0 [93.0 to 99.4]

2. Secondary Outcome: Percentage of Participants With On-treatment HCV Virologic Failure
Description: On-treatment HCV virologic failure was defined as one of the following:
  * Confirmed hepatitis C virus ribonucleic acid (HCV RNA) ≥ 100 IU/mL after HCV RNA < 15 IU/mL at any time point during treatment; or
  * Confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) during study drug treatment; or
  * HCV RNA ≥ 15 IU/mL at the end of treatment with at least 6 weeks of treatment.
Time Frame: 8 or 12 weeks (depending on treatment regimen)
Population: All enrolled participants who received at least 1 dose of study drug. Data are reported for the overall study population according to the prespecified analysis plan for this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: GLE/PIB for 8 or 12 weeks
Arm/Group | All Participants
Number analyzed (Participants) | 100
percentage of participants | 0 [0.0 to 3.7]

3. Secondary Outcome: Percentage of Participants With Post-treatment HCV Virologic Relapse
Description: Post-treatment HCV virologic relapse was defined as confirmed HCV RNA ≥ 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment as planned with HCV RNA levels < 15 IU/mL at the end of treatment and had post-treatment HCV RNA data; participants who had been shown to be re-infected were not considered to have relapsed.
Time Frame: From the end of treatment (8 or 12 weeks depending on treatment regimen) through 12 weeks after the last dose of study drug
Population: All enrolled participants who received at least 1 dose of study drug and who completed treatment, had HCV RNA < 15 IU/mL at final treatment visit, and had at least one post-treatment HCV RNA value. Data are reported for the overall study population according to the prespecified analysis plan for this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 100
percentage of participants | 1.0 [0.2 to 5.4]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug.
Description: Adverse events are reported for the overall study population according to the prespecified analysis plan for this study.
Groups:
- All Participants: All enrolled participants who received at least one dose of study drug.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 4/100
Other Adverse Events (participants affected / at risk) | 30/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=100)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=100)
NAUSEA (Gastrointestinal disorders) | 6 (6)
FATIGUE (General disorders) | 5 (5)
HEADACHE (Nervous system disorders) | 18 (18)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03219216/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT03219216/SAP_001.pdf